CLINICAL TRIAL: NCT05230641
Title: Cardiac Autonomic Dysfunction and Perioperative Outcomes After Neurosurgery
Brief Title: Cardiac Autonomic Dysfunction and Perioperative Outcomes
Acronym: CADPONS
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Collaborators: Vision Group on Science and Technology (Unknown); DyAnsys, Inc. (Industry)
Responsible Party: Principal Investigator, RP Sangeetha, Dr., National Institute of Mental Health and Neuro Sciences, India
Other Study IDs: NIMHANS/33 IEC(BS&NS DIV)/2021
Record Dates: First submitted 2022-01-12; First posted 2022-02-09 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Neurosurgical Patients
Keywords: cardiac dysautonomia; neurosurgery; heart rate variability; hypotension; anesthesia; major adverse cardiac events; perioperative outcome
MeSH Terms: conditions — Hypotension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is a prospective observational study
  Other Names: No interventions

SUMMARY:
The autonomic nervous system (ANS) is cardinal for maintaining systemic homeostasis and is pivotal for the baseline regulation and modulation of vital cardiovascular, hemodynamic, respiratory, gastrointestinal, and body temperature regulating functions. Pathological perturbations of the ANS leading to cardiac dysautonomia (CAD) affect one in 1000 population. Autonomic dysfunction can occur from a variety of pathological conditions such as ischemic heart disease, systemic hypertension, diabetes mellitus, neurological illnesses, neurotrauma, and cervical spine diseases. When patients with dysautonomia present for surgical procedures, they may manifest severe hemodynamic responses that may be less responsive to pharmacological interventions. Pre-existing autonomic dysfunction accentuates perioperative hemodynamic fluctuations during stressful events like direct laryngoscopy, endotracheal intubation, and extubation, and can result in major adverse cardiac events (MACE). The complications arising from CAD can prolong the duration of hospital stay and contribute to morbidity and mortality. Preoperative diagnosis of CAD helps in anticipation of and preparation for potentially severe adverse events in the perioperative period. Most neurosurgical patients are not candidates for detailed ANS examination in the supine and standing positions due to their underlying neurological condition. Real-time assessment of heart rate variability (HRV) using the ANSiscope equipment provides information on the sympathovagal balance during the immediate preoperative period and aids in the simple rapid bedside assessment of CAD. This study aims to examine the incidence of CAD through HRV assessment in neurosurgical patients, identify the potential risk factors for CAD in this population, and evaluate the impact of CAD on perioperative outcomes.

DETAILED DESCRIPTION:
Demographic and baseline clinical data including comorbid conditions and medication history will be collected. Baseline hemodynamic parameters - heart rate (HR) and systolic, diastolic, and mean blood pressure (SBP, DBP, MAP), rate pressure product (RPP) calculated as the product of HR and SBP and ANSindex (which informs the degree of dysautonomia and is derived noninvasively from a recording of 572 R wave to R wave intervals on an electrocardiogram) will be recorded in the immediate preoperative period.

Assessment of risk factors for preoperative CAD The investigators will explore potential risk factors for CAD in neurosurgical patients. The investigators postulate some known factors such as anxiety which will be diagnosed using the Visual analog scale for anxiety (VAS-A), age, gender, neurosurgical pathology, site-specific surgery (high cervical pathology, structural brain lesions, brainstem lesion, etc.), pre-existing diabetes mellitus and hypertension, and medications used for their treatment, higher American Society of Anesthesiology (ASA) grade, etc. to be associated with CAD in neurosurgical patients.

The investigators will explore the association between CAD and perioperative outcomes. Major Adverse Cardiac Events during Intra and postoperative period, in-hospital mortality, and duration of postoperative ICU and hospital stay.

Anesthesia will be administered as per the existing practice. Hemodynamic parameters HR, SBP, DBP, MAP at following time points - before and 1 and 2 min after induction of general anesthesia, before and at 1, 3, and 5 mins after tracheal intubation, and before and at 1, 3, and 5 mins after skull pin application, where applicable. Adverse hemodynamic events - persistent hypotension, arrhythmias, myocardial ischemia, cardiac failure, cardiac arrest) during the early (after anesthetic induction and before surgical incision), late (surgical incision to surgical closure) intraoperative period, recovery period (end of anesthesia to discharge from the operating room), post-anesthesia care unit (PACU) period (from arrival to discharge from PACU) and early postoperative period (up to 72 hours after surgery), neurological status (Glasgow Coma Scale) at hospital discharge, and duration of ICU and hospital stay will be recorded. The core temperature will be monitored during the intraoperative period to detect hypothermia (<35o C) or hyperthermia (>37.5 o C).

Sample size and statistical analysis Previous studies in the non-neurosurgical populations have determined the prevalence of CAD to vary from 25 to 73%. Considering an average prevalence of 50% in the neurosurgical population and a possible 5% margin of error, a sample size of 383 would be necessary for achieving a 95% confidence level. Hence the investigators plan to recruit 400 patients over a period of 1 year to account for potential dropouts from the study.

Data will be analyzed using Statistical Package for the Social Sciences (SPSS) or R software. Continuous variables will be compared by t-test, qualitative data by chi2 test, or Fisher exact test. Logistic regression will be used to identify the risk factors for cardiac autonomic dysfunction. A p < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80 years
* belonging to ASA grade 1-4
* scheduled for craniotomies or spinal surgeries under anesthesia

Exclusion Criteria:

* scheduled for redo procedures
* patients with preoperative arrhythmias and cardiac failure
* patients on preoperative inotropic support
* pregnant neurosurgical patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting patients scheduled for neurosurgical procedures at the National Institute of Mental Health and Neurosciences, Bengaluru will be recruited if they fulfill the study inclusion criteria during the period of study duration
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of cardiac autonomic dysfunction in neurosurgical patients | Before anesthesia administration for surgery
  To study the prevalence of cardiac autonomic dysfunction in neurosurgical patients

SECONDARY OUTCOMES:
Risk factors of cardiac autonomic dysfunction in neurosurgical patients | Baseline
  To identify risk factors of cardiac autonomic dysfunction in neurosurgical patients
Impact of cardiac autonomic dysfunction on hemodynamic stress response | During anesthesia procedure for surgery
  To assess the impact of cardiac autonomic dysfunction on hemodynamic stress response to laryngoscopy and intubation, anesthetic induction, and tracheal extubation
Impact of cardiac autonomic dysfunction on hemodynamic instability | During surgery
  To assess the impact of cardiac autonomic dysfunction on incidence, duration and severity of intraoperative hypotension and hypertension and requirement of pharmacological intervention
Impact of cardiac autonomic dysfunction on Major Adverse Cardiac Events | During and after surgery till discharge from the hospital, an average of 1 week
  To assess the impact of cardiac autonomic dysfunction on Major Adverse Cardiac Events namely, new onset myocardial ischemia, congestive cardiac failure, cardiac arrhythmias, cardiac arrest requiring resuscitation
Impact of cardiac autonomic dysfunction on temperature instability | During surgery
  To assess the impact of cardiac autonomic dysfunction on incidence of hypothermia and hyperthermia
Impact of cardiac autonomic dysfunction on duration of hospital stay | After surgery till the time of discharge from the hospital, an average of 1 week
  To assess the impact of cardiac autonomic dysfunction on duration of ICU and hospital stay
Impact of cardiac autonomic dysfunction on in-hospital mortality | After surgery till the time of discharge from the hospital, an average of 1 week
  To assess the impact of cardiac autonomic dysfunction on in-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha RP, Principal Investigator — National Institute of Mental Health and Neuro Sciences, India
Locations (1):
- NIMHANS hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be available with the Principal Investigator and shared with other researchers on request.

REFERENCES:
- [Background] Chakraborty T, Kramer CL, Wijdicks EFM, Rabinstein AA. Dysautonomia in Guillain-Barre Syndrome: Prevalence, Clinical Spectrum, and Outcomes. Neurocrit Care. 2020 Feb;32(1):113-120. doi: 10.1007/s12028-019-00781-w. PMID 31297663
- [Background] McGrane S, Atria NP, Barwise JA. Perioperative implications of the patient with autonomic dysfunction. Curr Opin Anaesthesiol. 2014 Jun;27(3):365-70. doi: 10.1097/ACO.0000000000000072. PMID 24722004
- [Background] Keyl C, Lemberger P, Palitzsch KD, Hochmuth K, Liebold A, Hobbhahn J. Cardiovascular autonomic dysfunction and hemodynamic response to anesthetic induction in patients with coronary artery disease and diabetes mellitus. Anesth Analg. 1999 May;88(5):985-91. doi: 10.1097/00000539-199905000-00004. PMID 10320156
- [Background] Polderman JAW, Sperna Weiland NH, Klaver MH, Biginski J, Horninge M, Hollmann MW, DeVries JH, Immink RV, Preckel B, Hermanides J. The prevalence of cardiovascular autonomic neuropathy and its influence on post induction hemodynamic variables in patients with and without diabetes; A prospective cohort study. PLoS One. 2018 Nov 26;13(11):e0207384. doi: 10.1371/journal.pone.0207384. eCollection 2018. PMID 30475825
- [Background] Hogan AM, Luck C, Woods S, Ortu A, Petkov S. The Effect of Orthostatic Hypotension Detected Pre-Operatively on Post-Operative Outcome. J Am Geriatr Soc. 2021 Mar;69(3):767-772. doi: 10.1111/jgs.16966. Epub 2020 Dec 11. PMID 33314116
- [Background] Mustafa HI, Fessel JP, Barwise J, Shannon JR, Raj SR, Diedrich A, Biaggioni I, Robertson D. Dysautonomia: perioperative implications. Anesthesiology. 2012 Jan;116(1):205-15. doi: 10.1097/ALN.0b013e31823db712. PMID 22143168
- [Background] Cheshire WP, Freeman R, Gibbons CH, Cortelli P, Wenning GK, Hilz MJ, Spies JM, Lipp A, Sandroni P, Wada N, Mano T, Kim HA, Kimpinski K, Iodice V, Idiaquez J, Thaisetthawatkul P, Coon EA, Low PA, Singer W. Corrigendum to "Electrodiagnostic assessment of the autonomic nervous system: A consensus statement endorsed by the American Autonomic Society, American Academy of Neurology, and the International Federation of Clinical Neurophysiology" [Clin. Neurophysiol. 132(2) (2021) 666-682]. Clin Neurophysiol. 2021 May;132(5):1194. doi: 10.1016/j.clinph.2021.02.006. Epub 2021 Mar 6. No abstract available. PMID 33685802
- [Background] Farbood A, Sahmeddini MA, Bayat S, Karami N. The effect of preoperative depression and anxiety on heart rate variability in women with breast cancer. Breast Cancer. 2020 Sep;27(5):912-918. doi: 10.1007/s12282-020-01087-y. Epub 2020 Apr 7. PMID 32266603
- [Background] Abhishekh HA, Nisarga P, Kisan R, Meghana A, Chandran S, Trichur Raju, Sathyaprabha TN. Influence of age and gender on autonomic regulation of heart. J Clin Monit Comput. 2013 Jun;27(3):259-64. doi: 10.1007/s10877-012-9424-3. Epub 2013 Jan 8. PMID 23297094
- [Background] Katsanos AH, Korantzopoulos P, Tsivgoulis G, Kyritsis AP, Kosmidou M, Giannopoulos S. Electrocardiographic abnormalities and cardiac arrhythmias in structural brain lesions. Int J Cardiol. 2013 Jul 31;167(2):328-34. doi: 10.1016/j.ijcard.2012.06.107. Epub 2012 Jul 16. PMID 22809542
- [Background] Ideguchi M, Kajiwara K, Yoshikawa K, Sadahiro H, Nomura S, Fujii M, Suzuki M. Characteristics of intraoperative abnormal hemodynamics during resection of an intra-fourth ventricular tumor located on the dorsal medulla oblongata. Neurol Med Chir (Tokyo). 2013;53(10):655-62. doi: 10.2176/nmc.oa2012-0401. Epub 2013 Sep 27. PMID 24077276
- [Background] Padley JR, Ben-Menachem E. Low pre-operative heart rate variability and complexity are associated with hypotension after anesthesia induction in major abdominal surgery. J Clin Monit Comput. 2018 Apr;32(2):245-252. doi: 10.1007/s10877-017-0012-4. Epub 2017 Mar 14. PMID 28293808
- [Background] Knuttgen D, Weidemann D, Doehn M. Diabetic autonomic neuropathy: abnormal cardiovascular reactions under general anesthesia. Klin Wochenschr. 1990 Dec 4;68(23):1168-72. doi: 10.1007/BF01815272. PMID 2280579